CLINICAL TRIAL: NCT06019325
Title: The Effect of Single Shot Rhomboid Intercostal Plane Block on Chronic Pain Incidence and Acute Pain Scores After Mastectomy Surgery
Brief Title: Rhomboid Intercostal Plane Block on Chronic Pain Incidence and Acute Pain Scores After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Başak Altıparmak, Associated Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 230022
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Postoperative Pain, Acute; Postoperative Pain, Chronic; Neuropathic Pain
Keywords: analgesia; acute pain; chronic pain; neuropathic pain; rhomboid intercostal block
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Neuralgia; Agnosia; Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients will be under general anesthesia and will not be aware if they receive a block procedure or not.
  The investigator, the data collector and the outcome assessor will be completely blind to the study groups. Only the care provider who will perform the block procedures will know the study groups, but she will not involve in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): After endotracheal intubation, patients will be positioned in lateral decubitus position. A linear ultrasound probe will be placed at the edge of scapula at the level of T5-T6. Under sterile conditions, the landmark points (rhomboid major muscle, 5th and 6th ribs, and intercostal muscles) will be observed and a block needle will be directed to the interfacial plane between rhomboid major muscle and intercostal muscle. RIB will be performed by injecting 30 ml of bupivacaine 0.25%.
  Interventions: Procedure: RIB
- Control Group (No Intervention): No block procedure will be performed in this group.

INTERVENTIONS:
Procedure: RIB — After endotracheal intubation, patients will be positioned in lateral decubitus position. A RIB will be performed at the level of T5-T6 by ultrasound guidance. A single shot block will be performed by injecting 30 ml of 0.25% bupivacaine to the interfacial plane between rhomboid major muscle and intercostal muscle.
  Arms: Study Group

SUMMARY:
Rhomboid intercostal block is used to block lateral cutaneous branches of intercostal nerves between T3 and T9 dermatomes. RIB has been reported to be successful in attenuating acute pain following breast surgeries. However, it's effect on chronic pain has not been evaluated yet. The primary hypothesis of the study is that the incidence of chronic pain of the patients who will receive Rhomboid intercostal block (RIB) following breast cancer surgery will be lower than the patients who will receive no block intervention at the postoperative 3rd month. The secondary hypothesis is that the incidence ofchronic pain of the patients who will receive Rhomboid intercostal block (RIB) following breast cancer surgery will be lower than the patients who will receive no block intervention at the postoperative 6th month. An other secondary hypothesis is that the total BPI-SF scores will be lower in the RIB group than control group at the postoperative 3rd and the 6th months.

DETAILED DESCRIPTION:
The study is designed as a prospective, double-blinded, randomize controlled study. The patients who will undergo mastectomy surgery with or without axillary dissection will be included in the study. Anesthesia will be inducted with intravenous (iv) thiopental 5 mg/kg, fentanyl 2 mcg/kg and rocuronium bromide 0.6 mg/kg. Following intubation, patients will be allocated into two groups according to a randomization table created by a professional statistician. In the study group, patients will receive a single shot Rhomboid Intercostal Block (RIB) with 30 milliliters of %0.25 bupivacaine and in the control group no block procedure will be performed. All patients will receive a standard analgesia protocol which will include an intraoperative intravenous (iv) infusion of dexketoprofen 50 mg and iv tramadol 1 mg/kg 15 minutes prior to the end of the surgery. Postoperative pain intensity of the patients will be evaluated by Numerical Rating Scale (NRS) which is a scale ranges between 0 (no pain) and 10 (the worst pain that a person can stand). Pain scores of the patients will be recorded at the postoperative 15. and 30. min in the recovery room and if the NRS score is 4 or more, iv fentanyl 1 mcg/kg will be applied. At the surgical ward, pain scores will be evaluated at the postoperative 1st, 2nd, 6th, 12th and 24th hours and if the NRS score is 4 or more, iv tramadol 50 mg will be applied as rescue analgesia. Opioid consumptions of the patients will be recorded at the postoperative 24th hour. At the postoperative 3. and 6. months, a pain doctor will evaluate all patients by using Brief Pain Inventory Short Form (BPI-SF) and Douleur Neuropathique 4 (DN4) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* Female
* Ages between 18-65
* Patients who will receive breast cancer surgery under general anesthesia

Exclusion Criteria:

* Alcohol or substance or chronic opioid consumption story
* Any pain killers intake in the last 24 hours prior to surgery
* Body mass index over 35 kg/m2
* Infection at the injection sites
* Known allergy to local anesthetics
* Known psychiatric diseases which prevents communication
* Operations longer than 3 hours

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
3rd month chronic pain | At the postoperative 3. month
  The presence of chronic pain will be evaluated by using the 5. question of Brief Pain Inventory Short Form at the postoperative 3rd month. The question ranges from 0 (which means no pain) to 10 points (which means worst pain). The score equal to or over 4 points indicates the presence of chronic pain. Primary outcome of the study is the difference in the incidence of chronic pain between study and control groups at the postoperative 3rd month.

SECONDARY OUTCOMES:
6th month chronic pain | At the postoperative 6. month
  The presence of chronic pain will be evaluated by using the 5. question of Brief Pain Inventory Short Form at the postoperative 6th month. The question ranges from 0 (which means no pain) to 10 points (which means worst pain). The score equal to or over 4 points indicates the presence of chronic pain. Secondary outcome of the study is the difference in the incidence of chronic pain between study and control groups at the postoperative 6th month.
3rd month total Brief Pain Inventory Short Form Score | At the postoperative 3. month
  Total score of Brief Pain Inventory Short Form of all patients will be recorded at the postoperative 3rd month. The form ranges from 0 point (best score) to 120 (worst score) points. The 3rd outcome of the study is the difference in total Brief Pain Inventory Short Form scores of patients in the study and control groups at the postoperative 3rd month.
6th month total Brief Pain Inventory Short Form Score | At the postoperative 6. month
  Total score of Brief Pain Inventory Short Form of all patients will be recorded at the postoperative 6th month. The form ranges from 0 point (best score) to 120 (worst score) points. The 3rd outcome of the study is the difference in total Brief Pain Inventory Short Form scores of patients in the study and control groups at the postoperative 6th month.
3rd month neuropathic pain | At the postoperative 3. month
  The presence of neuropathic pain which will be evaluated by using Douleur Neuropathique 4 (DN4) which ranges from 0 point (no pain) to 10 points (worst pain). Score equal to or over 4 points indicates the presence of neuropathic pain. The 5th outcome of the study is the difference in the incidence of neuropathic pain between the study and control groups.
6th month neuropathic pain | At the postoperative 6. month
  The presence of neuropathic pain which will be evaluated by using Douleur Neuropathique 4 (DN4) which ranges from 0 point (no pain) to 10 points (worst pain). Score equal to or over 4 points indicates the presence of neuropathic pain. The 6th outcome of the study is the difference in the incidence of neuropathic pain between the study and control groups at the postoperative 6th month.
acute pain | Postoperative 15. minute, 30. minute, 1.hour, 2nd hour, 6th hour, 12th hour, 24th hour
  Postoperative acute pain of the patients will be evaluated by using Numerical Rating Scale which ranges between 0 point (no pain) and 10 points (worst pain). The 7th outcome of the study is the difference in numerical rating scale scores between study and control groups.
opioid consumption | Postoperative 24th hour.
  Total opioid consumption of the patients will be recorded at the postoperative 24. hour.

CONTACTS AND LOCATIONS:
Overall Officials: BAKİYE UĞUR, Study Chair — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Training and Research Hospital, Muğla, MENTEŞE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with anyone